CLINICAL TRIAL: NCT00551447
Title: A Comparison of Treatment With Ezetimibe (SCH 58235) and Simvastatin Coadministration Versus Simvastatin in Attaining the National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) III Coronary Heart Disease (CHD) or CHD Risk Equivalent Strata Low-Density Lipoprotein Cholesterol (LDL-c)
Brief Title: A Study Comparing Ezetimibe Plus Simvastatin Versus Simvastatin Alone in Patients at Risk for Heart Disease (0653-023)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-023; MK0653-023; 2006_555
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Ezetimibe; Duration of Therapy; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe / Duration of Treatment: 27 Weeks
Drug: MK0733, simvastatin / Duration of Treatment: 27 Weeks
Drug: Comparator: simvastatin / Duration of Treatment: 27 Weeks

SUMMARY:
This purpose of this study is to determine if the administration of ezetimibe and simvastatin together is more effective than simvastatin alone in lowering LDL-C levels to a goal of <100 mg/dL in patients at risk for Heart Disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 at risk for Heart Disease who have LDL-C levels greater than or equal to 130 mg/dL and triglyceride level less than or equal to 350 mg/dL
* Patients must be able to maintain the National Cholesterol Education Program diet throughout the course of the study

Exclusion Criteria:

* Patients are excluded from the study if their weight is less than 50% of ideal body weight, if they are pregnant or lactating, have congestive heart failure, uncontrolled heart rhythm problems or a recent heart attack, coronary artery bypass surgery, or angioplasty. Additionally, patients with poorly controlled Type 1 or 2 diabetes mellitus, kidney disease, uncontrolled endocrine or metabolic disease, are known HIV positive, and uncontrolled high blood pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2002-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
LDL-C measurement (target goal = <100 mg/dL) | 27 Weeks

SECONDARY OUTCOMES:
Well tolerated in patients | 27 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] McKenney J, Ballantyne CM, Feldman TA, Brady WE, Shah A, Davies MJ, Palmisano J, Mitchel YB. LDL-C goal attainment with ezetimibe plus simvastatin coadministration vs atorvastatin or simvastatin monotherapy in patients at high risk of CHD. MedGenMed. 2005 Jul 14;7(3):3. PMID 16369229
- [Background] Feldman T, Koren M, Insull W Jr, McKenney J, Schrott H, Lewin A, Shah S, Sidisin M, Cho M, Kush D, Mitchel Y. Treatment of high-risk patients with ezetimibe plus simvastatin co-administration versus simvastatin alone to attain National Cholesterol Education Program Adult Treatment Panel III low-density lipoprotein cholesterol goals. Am J Cardiol. 2004 Jun 15;93(12):1481-6. doi: 10.1016/j.amjcard.2004.02.059. PMID 15194017
- [Background] Catapano A, Brady WE, King TR, Palmisano J. Lipid altering-efficacy of ezetimibe co-administered with simvastatin compared with rosuvastatin: a meta-analysis of pooled data from 14 clinical trials. Curr Med Res Opin. 2005 Jul;21(7):1123-30. doi: 10.1185/030079905X50642. PMID 16004682